CLINICAL TRIAL: NCT04158596
Title: Randomised, Double-blind, Multi-centre, Clinical Trial to Assess the Safety and Efficacy of SDX-3101, an Innovative Vibration Therapy Portable Device for the Treatment of Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP) in Adult Patients
Brief Title: Safety and Efficacy of SDX-3101 for the Treatment of Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Acronym: SDX-3101
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: SynDermix AG (Industry)
Collaborators: ISS AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDX-3101
Record Dates: First submitted 2019-11-05; First posted 2019-11-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The applied therapeutic vibrations generated by an acoustic coil have a defined sweeping frequency range.
  Interventions: Device: Vibration Therapy
- Control (Active Comparator): A control device with a different vibration pattern will be used as comparator intervention
  Interventions: Device: Vibration Therapy

INTERVENTIONS:
Device: Vibration Therapy — SDX-3101 is used for drug-free treatment of CRSsNP in adults.

SUMMARY:
The purpose of this clinical trial is to assess the safety and efficacy of SDX-3101 for treatment of adult patients with chronic rhinosinusitis without nasal polyps (CRSsNP) by investigating a vibration pattern of SDX-3101 compared to a control

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a common disease (e.g. 11% of adults in the UK report symptoms of CRS) leading to substantial health and socioeconomic burden with estimated healthcare costs in the USA of $772/patient/year (2011).

CRS is characterised by the long-term presence of multiple symptoms including facial pain/pressure in about 80% of CRS patients. Factors contributing to the pathophysiology of adult CRS include allergies, bacterial biofilms, asthma and exposure to various environmental pollutants. Computed tomography (CT) scans are often used to identify mucosal thickening and to identify any comorbid factors such as anatomic abnormalities.

It is known from the literature that low vibration frequency can improve blood flow, significantly reduce inflammation, and increase the fibroblast activity [13]. Therefore, SynDermix AG created the innovative high-technology, portable medical device SDX-3101 targeting a disease with high unmet medical need. The device offers a drug-free or eventually an add on treatment complying with the maximum demands of safety for the patients potentially avoiding undesirable drug effects or surgery. SDX-3101 is indicated for treatment of CRSsNP in adults

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects between 18 and 70 years old
* Diagnosed history of chronic rhinosinusitis without nasal polyps (CRSsNP) defined as per EPOS Guidelines.
* Moderate to severe baseline SNOT-20 GAV score (> 20)
* Willingness to stop nasal saline irrigation and drug therapy for CRSsNP (restart later on possible)

Exclusion Criteria:

* Subjects with local pathology that would compromise the ability to either administer the device or assess the benefits/risks (e.g. mucocele, antrochoanal polyp, facial trauma, radiation injury, or birth defect)
* Systemic corticosteroids if not stop for 14 days before study enrolment
* Subjects suffering from insufficiently controlled asthma
* Subjects suffering from insufficiently controlled allergic rhinitis (AR)
* Subjects with prior sinus operations within the last 4 months
* Subjects with known primary ciliary dyskinesia/cystic fibrosis
* Subjects with serious underlying medical condition
* Ongoing oncological treatments
* Known hypersensitivity to materials in direct contact with the skin
* Metal or metal-like implant (incl. ceramic) located in the head or neck area. Unremovable hearing aids
* Patients with implanted cardiac pace-maker
* Women who are pregnant or breast feeding
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
SNOT-20 GAV | 12 weeks
  The primary endpoint is the change in subjective symptoms as quantified by the German validated disease-specific 20-item Sino-nasal Outcome Test (SNOT-20 GAV) after 12 weeks. Superiority is defined as more than minimal clinically important difference (MCID) of 8.9 points to active control of SNOT-20 score at 12 weeks.

SECONDARY OUTCOMES:
Lund-Kennedy Score | day 0, day 14, week 6, 12 and at 6, 9 and 12 months
  We use the Lund-Kennedy endoscopic scoring system to measure the patient's nasal cavity based on there were edema, vesicles, adhesions, scars and polyps
Overall disease control | day 14, week 6, 12 and at 6, 9 and 12 months
  Need for systemic medication, steroid or antibiotic, number of days
Need for surgical intervention | day 14, week 6, 12 and at 6, 9 and 12 months
  Capture surgical intervention
Ability to perform normal activities | day 0, day 14, week 6, 12 and at 6, 9 and 12 months,
  Measured with the SNOT-20 GAV
Acceptability of treatment | day 14, week 6, 12 and at 6, 9 and 12 months
  Measurement of Visual Analogue Scale 0 to 5, 0 is unacceptable to 5 fully accepted
Overall score SNOT-20 | day 0, day 14, week 6, 12 and at 6, 9 and 12 months
  The SNOT-20 has a maximum score of 100 and a minimum score of 0. Higher values represent a worse outcome
Pain in the face | day 0, day 14, week 6, 12 and at 6, 9 and 12 months
  Measured on a 4-point scale, (0=no symptoms; 1=mild symptoms present, but not troublesome; 2=moderate symptoms that were frequently troublesome but not sufficiently so to interfere with normal daily activities or sleep; 3=severe symptoms that interfered with normal daily activities or sleep)
Global impression by investigator | day 0, week 6, 12 and at 12 months,
  Measured with Visual Analogue Scale 0 to 10, 0 is unsatisfactory 10 is optimal outcome

OTHER OUTCOMES:
Saccharine test | day 0, week 6, 12 weeks and at 12 months
  Evaluate muco-ciliary clearance time
Reduction in inflammatory markers | day 0, day 14, week 6, 12
  Assessed by Biomarkers: IL-1β, IL-2, IL-4, IL-10, IL-12 and IgE in nasal secretion
Exhaled nasal Nitric Oxide (nNO) levels | day 0, day 14, week 6, 12 and 12 months
  only in a subpopulation in selected site/s

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Camozzi, MD, Study Director — SynDermix AG
Locations (8):
- Kardinal Schwarzenberg Klinikum GmbH, Schwarzach im Pongau, Austria
- Germany (5):
  - Praxis Dr.med. Decot, Dreieich
  - ENT Research Institut für Klinische Studien, Essen
  - HNO Praxis am Neckar, Heidelberg
  - HNO - Arzt Allergologe Studienzentrum, Viernheim
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Switzerland (2):
  - Universitätsklinik für Hals-, Nasen- und Ohrenkrankheiten, Kopf- und Halschirurgie, Inselspital,, Bern
  - Department of ENT, Head and Neck Surgery Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No